CLINICAL TRIAL: NCT02542579
Title: Composition of Gastric and Duodenal Microbiota in Dyspeptic Subjects
Brief Title: Gastric and Duodenal Microbiota in Dyspeptic Subjects
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Sun-Young Lee, Professor, Konkuk University Medical Center
Other Study IDs: KUH1010691
Record Dates: First submitted 2015-08-23; First posted 2015-09-07 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Microbial Colonization; Gastritis
Keywords: Helicobacter pylori; Dyspepsia
MeSH Terms: conditions — Communicable Diseases; Gastritis; Dyspepsia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gastric and duodenal mucosa
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Subjects for pyrosequencing analysis: Dyspeptic subjects who visited for evaluation and agreed on 16S rRNA pyrosequencing analysis
  Interventions: Genetic: 16S rRNA pyrosequencing analysis

INTERVENTIONS:
Genetic: 16S rRNA pyrosequencing analysis — Next generation sequencing analysis will be done for 16S rRNA V1,2 hypervariable regions at Biocore (Seoul, Korea).

SUMMARY:
The composition of gastric microbiota is determined by the status of Helicobacter pylori infection. In subjects who have never been infected by H. pylori, gastric microbiota includes various bacteria, creating ideal microbial diversity. This ideal microbial diversity is destroyed by H. pylori infection at low intragastric pH. Since it is difficult for most bacteria to proliferate within an acidic stomach, relative H. pylori abundance gives rise to microbial dysbiosis. Conversely, unideal microbial diversity is often observed in infected individuals with impaired gastric secretory ability at hypochlorhydric condition. Bacteria producing carcinogenic N-nitrosamine compounds are often detected in individuals with past or chronic H. pylori infection at high intragastric pH. Nonetheless, microbial imbalance that occurs in the earlier phase before gastric carcinognenesis is uncertain.

DETAILED DESCRIPTION:
Dominant colonization of a specific microbiota leading to dysbiosis may lead to inflammation of the mucosa. We hypothesized that the degree of inflammation depend on the composition of microbiota. This study was aimed to define gastric and duodenal microbiota leading to abnormal histopathology. We further tried to elucidate whether the composition of duodenal microbiota is altered by gastric microbiota.

Among the dyspeptic subjects who visited for upper gastrointestinal (UGI) endoscopy, subjects with drug intake (antibiotics, PPIs, laxatives, antidepressants, statins, metformin) within 3 months will be excluded. Three biopsies will performed at the greater curvature side of the mid-antrum, greater curvature side of the mid-body, and at the duodenum, respectively. Next generation sequencing analysis will be performed for 16S rRNA variable regions using the biopsied samples.

Primary study endpoint is 16S rRNA sequencing findings of gastric and duodenal microbiota.

Secondary endpoints are microbiota linked with higher degrees of inflammation, activity, atrophy and intestinal metaplasia based on the updated Sydney classification. Furthermore, correlation between the microbiota and endoscopy finding will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Dyspeptic subjects who visited for evaluation including upper gastrointestinal endoscopy and biopsies
* Age >20 years old

Exclusion Criteria:

* Underlying disease(s) that requires managements
* Recent intake of drug(s)
* History of gastrectomy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dyspeptic subjects for analysis
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Next generation sequencing analysis for microbiota | up to 6 months
  16S rRNA pyrosequencing analysis findings of the gastric and duodenal biopsies

SECONDARY OUTCOMES:
Updated Sydney classification | up to 6 months
  0=none, 1=mild, 2= moderate, 3=marked infiltration
Gastrointestinal endoscopy finding | up to 6 months
  Upper gastrointestinal endoscopy findings
Gastrointestinal symptom and food intake score | up to 6 months
  Scoring system published in Neurogastroenterol Motil 2016;28:1401-1408

CONTACTS AND LOCATIONS:
Overall Officials: Sun-Young Lee, M.D., Ph.D., Principal Investigator — Konkuk University
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SY, Moon HW, Hur M, Yun YM. Validation of western Helicobacter pylori IgG antibody assays in Korean adults. J Med Microbiol. 2015 May;64(Pt 5):513-518. doi: 10.1099/jmm.0.000050. Epub 2015 Mar 9. PMID 25752852
- [Background] Lee SP, Lee SY, Kim JH, Sung IK, Park HS, Shim CS, Moon HW. Correlation between Helicobacter pylori infection, IgE hypersensitivity, and allergic disease in Korean adults. Helicobacter. 2015 Feb;20(1):49-55. doi: 10.1111/hel.12173. Epub 2014 Sep 25. PMID 25257099
- [Background] Lee SY. Future candidates for indications of Helicobacter pylori eradication: do the indications need to be revised? J Gastroenterol Hepatol. 2012 Feb;27(2):200-11. doi: 10.1111/j.1440-1746.2011.06961.x. PMID 22098099